CLINICAL TRIAL: NCT07055269
Title: Assessment of Liver Metabolic Alterations in Vivo in Patients With Citrin Deficiency and Healthy Subjects by Metabolic Labeling With Stable Isotopes
Brief Title: Liver Metabolic Functions in Patients With Citrin Deficiency and Healthy Subjects
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Haeberle (Other)
Collaborators: Citrin Foundation (Unknown); Marc Hellerstein, University of Berkeley (Unknown)
Responsible Party: Sponsor-Investigator, Johannes Haeberle, Head of Metabolic Laboratory, University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-00730
Record Dates: First submitted 2025-06-25; First posted 2025-07-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Citrin Deficiency
Keywords: Citrin Deficiency; Adolescent and Adult Citrin Deficiency, AACD; SLC25A13; liver metabolic flux; ureagenesis; Citrin
MeSH Terms: conditions — Adult-onset citrullinemia type 2

STUDY DESIGN:
Intervention Model Description: Cross-sectional observational study, non-randomised
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AACD patient (Experimental): isotope tracer for ureagenesis and liver metabolic flux
  Interventions: Other: liver metabolic flux; Other: ureagenesis capacity
- healthy volunteer (Experimental): isotope tracer for ureagenesis and liver metabolic flux
  Interventions: Other: liver metabolic flux

INTERVENTIONS:
Other: liver metabolic flux — All participants will be given heavy water (2H2O, deuterium-labelled) and [U-13C6]-fructose orally, each followed by the collection of one blood plasma sample. Additional biochemical and clinical parameters including liver fat content by MRI, liver fibrosis and cirrhosis by ultrasound imaging and plasma biochemical profiles will be analyzed.
Other: ureagenesis capacity — urea and urea cycle metabolites and their enrichment after oral administration of a stable isotope tracer 15NH4Cl will be measured to examine the liver's ability to detoxify ammonia.
  Arms: AACD patient

SUMMARY:
Citrin is an aspartate-glutamate transporter in the liver that facilitates the urea cycle pathway for ammonia detoxification via ureagenesis. It is also thought to be involved in liver energy metabolism as a component of the malate-aspartate shuttle. The clinical presentation in patients supports the hypothesis that liver glycolytic, gluconeogenic and lipogenic functions are compromised in citrin deficiency, but none of the key hepatic pathway fluxes have been measured in patients to date. This is the first study that will examine the liver metabolic fluxes in patients with citrin deficiency.

Liver metabolic functions will be examined by metabolic flux assays and biochemical measurements after application of stable isotopes 2H2O and [U-13C6]-fructose. Urea cycle metabolites and their enrichment after application of a stable isotope tracer 15NH4Cl will be measured to examine the liver's ability to detoxify ammonia into urea.

ELIGIBILITY:
Inclusion criteria for AACD patients are:

* Subjects with citrin deficiency, confirmed by genetic analysis to carry pathogenic variant(s) in the SLC25A13 gene
* Age from 18 years to 65 years inclusive
* Male or female
* Written informed consent has been given
* Understands and is willing, able and likely to comply with study procedures and restrictions

Inclusion criteria for healthy subjects are:

* Age from 18 years to 65 years inclusive, and not more than five years younger or older than the specified paired participant from the AACD group
* Same sex as the specified paired participant from the AACD group
* Same ethnicity the specified paired participant from the AACD group
* Written informed consent has been given
* Understands and is willing, able and likely to comply with study procedures and restrictions

Exclusion criteria for AACD patients are:

* acute and chronic disease requiring treatment of any kind, other than his/her AACD
* females who are pregnant or lactating or attempting to become pregnant
* use of any medication which, in the opinion of the investigator, is likely to interfere with liver function

Exclusion criteria for healthy subjects are:

* carry any pathogenic variant in the SLC25A13 gene
* current or recurrent disease that could affect the metabolic function of the liver
* acute and chronic disease requiring treatment of any kind
* females who are pregnant or lactating or attempting to become pregnant
* use of any medication which, in the opinion of the investigator, is likely to interfere with liver function
* weight loss ≥10% within 3 months before study screening
* daily alcohol consumption of more than 2 standard-sized beer for men and more than 1 standard-sized beer for women, or the equivalent
* BMI > 30 kg/m2
* currently smoking >1 cigarette daily
* liver transplant recipients
* type 1 and 2 diabetes
* currently on a ketogenic diet
* currently taking medium chain triglyceride (MCT) supplements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Liver metabolic flux | 5 days
  Liver metabolic flux will be measured by assessing the distribution of the administered isotope tracers [U-13C6]-fructose and heavy water.

SECONDARY OUTCOMES:
Ureagenesis capacity | 1 day
  Patients will receive an oral dose of 2 mg/kg of the 15NH4Cl tracer diluted in water. Blood will be collected at various time points up to 2 hours after tracer administration to assess the body's ability to remove ammonia.
adverse events | 5 days
  Safety and tolerability of 2H2O, [U-13C6]-fructose and 15NH4Cl
liver fat content | 1 day
  Magnetic resonance imaging of the liver for fat content
Liver fibrosis | 1 day
  Ultrasound imaging of the liver to assess fibrosis and cirrhosis
Clinical symptoms | 1 day
  Clinical presentation and fatigue will be measured through questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- University Children's Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No